CLINICAL TRIAL: NCT04298008
Title: Combination of AZD6738 Plus Durvalumab in Refractory Biliary Tract Cancer in Patients Who Have Failed Immunotherapy
Brief Title: AZD6738 Plus Durvalumab in Biliary Tract Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Do-Youn Oh, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTC-IO RR
Record Dates: First submitted 2020-02-25; First posted 2020-03-06 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Bile Duct Cancer; Chemotherapy Effect
MeSH Terms: conditions — Bile Duct Neoplasms | interventions — ceralasertib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD6738 + Durvalumab Cohort (Experimental): This is a study enrolling advanced BTC patients who have been previously treated with immunotherapy, to explore the combination of AZD6738+durvalumab
  Interventions: Drug: AZD6738; Drug: Durvalumab

INTERVENTIONS:
Drug: AZD6738 — AZD6738 (240 ) mg bid on D15-D28 Every 4 weeks
Drug: Durvalumab — Durvalumab 1500 mg iv on D1 Every 4 weeks

SUMMARY:
This trial will enroll advanced biliary tract cancer patients who have been previously treated with immunotherapy in either the 2nd or 3rd line.

Patients will be treated with AZD6738 and Durvalumab combination.

DETAILED DESCRIPTION:
This is a single arm, phase II study. Advanced BTC patients who have been previously treated with immunotherapy in either the 2nd or 3rd line will be enrolled.

Patients will be treated with AZD6738 and Durvalumab combination.

One cycle consists of 4weeks. Response evaluation will be done every 8 weeks (every 2 cycles) of treatment

1. Tumor biopsy is mandatory: screening, after 8weeks (1st-response evaluation), at disease progression (PD)
2. blood sampling for biomarker study is mandatory: every cycles
3. To evaluate the metabolic changes by AZD6738 and Durvalumab combination : 18 F-FDG PET is mandatory : screening, after 8 weeks (1st-response evaluation)

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and any locally-required authorization obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
2. Age > 20 years at time of study entry
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Life expectancy of > 16weeks
5. Histologically proven BTC, including intrahepatic cholangiocarcinoma, extrahepatic bile duct cancer, gallbladder cancer, ampulla of vater cancer
6. Unresectable or recurrent
7. Failed immunotherapy for their advanced BTC (the patient may have also received chemotherapy in the 1 or 2L)
8. At least one measurable lesion that can be accurately assessed at baseline by computed tomography (CT) (magnetic resonance imaging [MRI] where CT is contraindicated) and is suitable for repeated assessment as per RECIST 1.1.
9. Body weight >30kg
10. Adequate normal organ and marrow function measured within 28 days prior to administration of study treatment as defined below :

    * Haemoglobin ≥9.0 g/dL
    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    * Platelet count ≥ 100x 109/L
    * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). (This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.)
    * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
    * Patients must have creatinine clearance estimated of ≥51 mL/min using the Cockcroft-Gault equation or based on a 24 hour urine test :

    Estimated creatinine clearance = (140-age [years]) x weight (kg) (x F)a serum creatinine (mg/dL) x 72 a where F=0.85 for females and F=1 for males.
11. Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1.

Postmenopausal is defined as:

* Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
* Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50
* radiation-induced oophorectomy with last menses >1 year ago
* chemotherapy-induced menopause with >1 year interval since last menses
* surgical sterilisation (bilateral oophorectomy or hysterectomy) 12. Male patients must use a condom during treatment and for 6 months after the last dose of AZD6738 when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception ([see appendix H for acceptable methods]) if they are of childbearing potential 13. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 3 weeks
2. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
3. Any previous treatment with ATR inhibitor
4. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
5. Receipt of the last dose of anti-cancer therapy (chemotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) within 21 days of the first dose of study drug .2 The minimum washout period for immunotherapy is 42 days
6. Mean QT interval:

   Mean resting corrected QT interval (QTc) >470 msec for females and >450 for men, obtained from 3 electrocardiograms (ECGs) 2-5 minutes apart using the Fredericia formula

   - Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as congestive heart failure, unstable angina pectoris, acute myocardial infarction, hypokalaemia, congenital long QT syndrome, immediate family history of long QT syndrome or unexplained sudden death under 40 years of age, conduction abnormality not controlled with pacemaker or medication.
7. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. The following are exceptions to this criterion

   The following are exceptions to this criterion:
   * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
   * Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
   * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
8. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
9. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
10. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug
11. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.

    Patients must have recovered from any effects of any major surgery
12. History of allogenic organ transplantation.
13. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    * Patients with celiac disease controlled by diet alone
14. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
15. History of another primary malignancy except for

    * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease
16. History of leptomeningeal carcinomatosis
17. Brain metastases or spinal cord compression. Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
18. History of active primary immunodeficiency
19. Active infection or immunocompromised patients including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B , hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Subjects with simple HBV carrier, a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
20. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
21. Female patients who are pregnant or breastfeeding
22. Male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 6 months after the last dose of AZD6738 or durvalumab monotherapy. (including sperm donation for male patients)
23. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
24. Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.

    Concomitant use of known potent (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) inhibitors or CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting study treatment is five half-lives, except for St-Johns' wort, which is 3 weeks.
25. Diagnosis of ataxia telangiectasia.
26. Refractory nausea and vomiting, chronic gastrointestinal diseases or previous significant bowel resection, with clinically significant sequelae that would preclude adequate absorption of AZD6738.
27. Haematuria: +++ on microscopy or dipstick.
28. Hypotension (<100/60 mmHg) or clinically relevant orthostatic hypotension, including a fall in blood pressure of >20 mmHg.
29. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
disease control rate (DCR) of AZD6738 and Durvalumab combination | through study completion, an average of 1 year
  Disease control rate based on RECIST v1.1

SECONDARY OUTCOMES:
overall response rate (ORR) of AZD6738 and Durvalumab combination | through study completion, an average of 1 year
  overall response rate (ORR) based on RECIST v1.1
progression-free survival of AZD6738 and Durvalumab combination | through study completion, an average of 1 year
  Time from enroll until disease progression or death
duration of response of AZD6738 and Durvalumab combination | through study completion, an average of 1 year
  Time from documentation of tumor response to disease progression
overall survival of AZD6738 and Durvalumab combination | every 12 weeks until death or up to 5 years
  Time from enroll until death from any cause
Safety and tolerability as measured by number and grade of toxicity events | through study completion, an average of 1 year
  CTCAE v5.0
quality of life measurement | through study completion, an average of 1 year
  EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No